CLINICAL TRIAL: NCT05048732
Title: Imaging Apoptosis for Lymphoma Treatment Response
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Futility
Sponsor: Washington University School of Medicine (Other)
Collaborators: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Diagnostic
Other Study IDs: 202108112
Record Dates: First submitted 2021-09-08; First posted 2021-09-17 (Actual); Last update posted 2024-05-30 (Actual); Status verified 2024-05

CONDITIONS: Diffuse Large B Cell Lymphoma
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Cohort 1 = Healthy Volunteers (Experimental): * Healthy volunteers (N=6, three male, three female) will be recruited to undergo a single 18F-FAT PET/CT imaging session for radiation dosimetry estimates.
  * 18F-FAT administration followed by body imaging at 3 time points
    * 0-60 min = multiple quick body scans
    * 120 min post injection = body scan
    * 240 min post injection = body scan
  Interventions: Drug: 18F-FluorApoTrace
- Cohort 2a: Newly Diagnosed DLBCL patients being treated with R-CHOP (Experimental): -N= 6 : 18F-FAT imaging session at baseline and Day 2-4 following Cycle 1 standard of care therapy.
  Interventions: Drug: 18F-FluorApoTrace
- Cohort 2b: Newly Diagnosed DLBCL patients being treated with R-CHOP (Experimental): -N=9: 18F-FAT imaging session at baseline and best time point determined from Cohort 2a (2 days post Cycle 1 standard of care therapy)
  Interventions: Drug: 18F-FluorApoTrace

INTERVENTIONS:
Drug: 18F-FluorApoTrace — -The dose of 18F-FluorApoTrace to be given is 5 mCi
  Other Names: 18F-FAT

SUMMARY:
Apoptosis is a specific form of cell death that leads to clearance of dead cells without causing inflammation or injury to normal adjacent tissues. Targeted cancer therapeutics that target this pathway for tumor cell death induction are in development, but few specific biomarkers of apoptosis are available to assess treatment response. Apoptosis also occurs in response to standard anthracycline or combination therapies such as rituximab, cyclophosphamide, doxorubicin, vincristine, and prednisolone (R-CHOP), rituximab, etoposide, phosphate, prednisone, vincristine sulfacte, cyclophosphamide, and doxorubicin hydrocholoride (R-EPOCH) used to treat many different histopathological types of lymphoma including Hodgkin and non- Hodgkin lymphoma such as diffuse large B-cell lymphoma (DLBCL), Burkitts lymphoma, primary mediastinal B-cell lymphoma and double hit DLBCL. Caspase-3 activation occurs as a result of apoptosis and may be a specific marker of apoptosis. Therefore, this study will assess whether 18F-FluorApoTrace (18F-FAT), a caspase-3 targeted tracer, has a reasonable dosimetry profile and can be used to detect apoptosis in patients with lymphoma being treated with standard therapy.

ELIGIBILITY:
Inclusion Criteria (Healthy Volunteers):

* Adult 18 years of age or older
* No known hematological disorders
* Considered healthy based on assessment by Principal Investigator (PI).
* Able to provide informed consent
* Able to comprehend and willing to follow instructions for study procedures as called for by the protocol.
* Capable of lying still and supine within the PET/CT scanner for up to 1 hour at a time.

Exclusion Criteria (Healthy Volunteers):

* No illicit drug use or other inhaled drug use (including pharmacologic agents, recreational agents or illicit drugs) within the past year per self-reporting mechanisms.
* No history of claustrophobia or other preventing condition that has previously or would interfere with completion of protocol specified imaging sessions.
* Not currently pregnant or nursing: Subject must be surgically sterile (has had a documented bilateral oophorectomy and/or documented hysterectomy), postmenopausal (cessation of menses for more than 1 year), non-lactating, OR of childbearing potential for whom a urine pregnancy test (with the test performed within the 24 hour period immediately prior to administration of 18 F-FAT) is negative

Inclusion Criteria (Participants with Diffuse Large B Cell Lymphoma):

* Men or women 18 years of age or older with a new diagnosis of lymphoma who will be treated with standard of care therapy for curative intent and at least one measurable (RECIST 1.1), FDG-avid lesion. OR recurrent DLBLC with at least one measurable (RECIST 1.1) FDA-avid lesion and a minimum of 12 months since last receiving treatment.
* If applicable at least one FDG avid lesion accessible for biopsy (ultrasound guided preferred)
* Able to provide informed consent
* Able to tolerate standard of care systemic therapy as recommended by referring physician(s).

Exclusion Criteria (Participants with Diffuse Large B Cell Lymphoma):

* Not currently pregnant or nursing: Subject must be surgically sterile (has had a documented bilateral oophorectomy and/or documented hysterectomy), postmenopausal (cessation of menses for more than 1 year), non-lactating, OR of childbearing potential for whom a urine pregnancy test (with the test performed within the 24 hour period immediately prior to administration of 18 F-FAT) is negative
* Not currently enrolled in another study using an investigational drug

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2021-12-06 (Actual); Primary Completion 2024-02-10 (Actual); Study Completion 2024-02-10 (Actual)

PRIMARY OUTCOMES:
Whole body effective dose (in rems) of a 5 mCi injection of 18F-FAT (Cohort 1 only) | Day 1
  -The time activity curves will be created using all the scans obtained and integrated to determine organ residence times. This data, plus the counts and volumes from urine collection(s) after tracer injection, will then be used to calculate the dosimetry using OLINDA/EXM v1.1. The calculated residence times will be used with the program OLINDA/EXM for 18F and using the adult human (adult female or male) model to calculate the whole body effective dose.
Radiation doses (rems) to critical organs (Cohort 1 only) | Day 1
  The time activity curves will be created using all the scans obtained and integrated to determine organ residence times. This data, plus the counts and volumes from urine collection(s) after tracer injection, will then be used to calculate the dosimetry using OLINDA/EXM v1.1. The calculated residence times will be used with the program OLINDA/EXM for 18F and using the adult human (adult female or male) model to calculate the individual organ radiation dose.
Change in mean standard uptake value (SUV) (Cohort 2 only) | Through completion of early interim treatment monitoring scan (estimated to be 14 days)
  -30 minutes and 60-90 minutes post pre-treatment baseline monitoring scan and 30 minutes and 60-90 minutes post early interim treatment monitoring scan
Change in maximum standard uptake value (SUV) (Cohort 2 only) | Through completion of early interim treatment monitoring scan (estimated to be 14 days)
  -30 minutes and 6-90 minutes post pre-treatment baseline monitoring scan and 30 minutes and 60-90 minutes post early interim treatment monitoring scan

SECONDARY OUTCOMES:
Distribution volume ratio (DVR) (Cohort 2 only) | Through completion of early interim treatment monitoring scan (estimated to be 14 days)
  -DVR will be calculated by reference region Logan plot analysis, in the largest (by size) and most FDG-avid (by maximum SUV) lymphoma lesions.
Change in percent positive caspase-3 staining (Cohort 2 only) | Baseline and post-treatment (estimated to be 14 days)
  * Biopsy samples from baseline and post-treatment will be collected. Immunohistochemical analysis will be performed for caspase-3 staining.
  * The preference for the post-treatment biopsy is for the biopsy to be performed on the same day as 18F-FAT imaging with imaging occurring prior to biopsy (either 2 or 4 days after receiving cycle 1 of R-CHOP). However, due to scheduling conflicts biopsy performed 2-7 days after cycle 1 R-CHOP therapy will be allowed.
  * The staining intensity will be assessed semi-quantitatively using a four-point scale (No Signal=0, Mild=1, Moderate=2, Strong=3). The percentage of stained cells at each intensity level will also be graded typically as 0 (<5%), 1 (5-25%), 2 (26-50%), 3 (51-75%), and 4 (>75%). The intensity score and percentage of positive cells will be then added to produce the final scores (0-7).

CONTACTS AND LOCATIONS:
Overall Officials: Farrokh Dehdashti, M.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu